CLINICAL TRIAL: NCT04823312
Title: Early Feasibility Study: Evaluation of Medtronic Duo Extended Set With 670G Pump Therapy
Brief Title: Evaluation of Medtronic DUO Extended Set
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Atlanta Diabetes Associates (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ADA-001
Record Dates: First submitted 2021-03-18; First posted 2021-03-30 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Diabetes Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Medtronic Duo Extended Set (Experimental): These subjects will be using 4 Duo Extended sets that will serve as an exploratory pilot study to assess the 7-day survival of the Duo Extended set.
  Interventions: Device: Experimental prospective single arm evaluating the Medtronic Duo Extended Set

INTERVENTIONS:
Device: Experimental prospective single arm evaluating the Medtronic Duo Extended Set — Subjects will be using 4 Duo extended sets that will serve as an exploratory pilot study to assess the 7-day survival of the Duo Extended set.
  Other Names: Medtronic DUO Extended Set with 670G Pump Therapy

SUMMARY:
This study is a single-center, non-randomized, prospective single arm study of adult subjects with type 1 diabetes utilizing 670G insulin pump therapy with Continuous Glucose Monitoring (CGM). These subjects will be using 4 DUO Extended sets that will serve as an exploratory pilot study to assess the 7-day survival of the Duo Extended set.

DETAILED DESCRIPTION:
Up to 20 adult subjects will be enrolled at the research center. Atlanta Diabetes Associates (ADA), with at least 15 subjects meeting the eligibility criteria. Eligibility criteria will be assessed at the screening visit and confirmed prior to Visit 2. At Visit 2, subjects will be provided supplies, including the DUO device, and will be trained on insertion. Each subject will wear their own MiniMed 670G insulin system including Guardian sensor (new sensor with transmitter will be provided for the study) and a DUO Extended set. The infusion set in the DUO Extended will be used for insulin infusion and the sensor in the DUO Extended will be blinded with a specific recorder connected to each sensor.

Guardian Sensor (3) and the SMBG measurements will be used for making therapy decisions as approved for the 670G system. Subjects will upload their pump, Contour meter and GS3 sensor data each week, which will be reviewed by an investigator. Subjects will wear the DUO device for a total of four weeks. At Visit 6, subjects will come to the site to have devices uploaded, to return the investigational devices, to have a skin assessment and for labs to be drawn.

ELIGIBILITY:
Inclusion Criteria:

1. Has type 1 diabetes for more than one year.
2. Subject is on the MiniMed 670G insulin pump therapy within1 year prior to screening.
3. Subject is currently using Auto Mode at least 75% of the time and willing to utilize Auto Mode and Duo device during the study.
4. Subject is willing and able to perform study procedures as per investigator discretion.
5. Subject is willing to take one of the following two insulins: Humalog or Novolog

Exclusion Criteria:

1. Subject is actively participating in an investigational study (drug or device) wherein he/she has received treatment from an investigational study drug or investigational study device in the last 2 weeks.
2. Subject is female and has a positive pregnancy screening test.
3. Subject is female of childbearing age and who is sexually active should be excluded if she is not using a form of contraception deemed reliable by investigator.
4. Subject is female and plans to become pregnant during the study.
5. Subject has Glycosylated hemoglobin (HbA1c) > 8.5 % at time of screening.
6. Subject has had a history of 1 or more episodes of severe hypoglycemia.
7. Subject has taken any oral, injectable, or IV glucocorticoids within 8 weeks from time of screening visit, or plans to take any oral, injectable, or IV glucocorticoids during the course of the study.
8. Subject is unable to tolerate tape adhesive in the area of Duo™ Extended set or sensor.
9. Subject has any unresolved adverse skin condition, including infection, in the area of Duo™ Extended set or sensor placement (e.g., psoriasis, dermatitis herpetiformis, rash, Staphylococcus infection).
10. Subject has had Diabetic Ketoacidosis (DKA) in the 12 months prior to screening visit.
11. Subject is currently abusing illicit drugs.
12. Subject is currently abusing alcohol.
13. Subject has history of adrenal disorder.
14. Subject has a history of inpatient psychiatric treatment in the past 6 months prior to screening.
15. Subject has any condition that the Investigator believes would interfere with study participation.
16. Subject has a history of visual impairment which would not allow subject to participate in the study and perform all study procedures safely, as determined by the investigator.
17. Subject has a sickle cell disease, hemoglobinopathy; or has received red blood cell transfusion or erythropoietin within 3 months prior to time of screening.
18. Subject plans to receive red blood cell transfusion or erythropoietin over the course of study participation.
19. Subject is using pramlintide (Symlin), SGLT2 inhibitors, GLP agonists, biguanides, DPP-4 inhibitors or sulfonylureas more than 2 weeks from time of screening.
20. Subject has been diagnosed with chronic kidney disease, having an estimated glomerular filtration rate (eGFR)< 60mL/min/1.73 m2, requiring dialysis, or resulting in chronic anemia.
21. Subject has history of cardiovascular disease defined as any ischemic related event or clinically significant arrythmia.
22. Subject has hypothyroidism and has out of reference range thyroid-stimulating hormone (TSH) on screening visit.
23. Subject plans to have medical imagining (e.g., MRI, diathermy services, CT scans, etc.) over the course of the study.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-03-18 (Actual); Primary Completion 2021-10-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Number of subjects with Duo Extended set failures due to unexplained hyperglycemia (i.e. suspected occlusion) at the end of Day 7. | 7 days
  Unexplained hyperglycemia

SECONDARY OUTCOMES:
Number of subjects with a rate of infusion set survival of 7 days or greater, excluding those that kinked on insertion or accidentally pulled out. | 7 days
  Infusion set survival

CONTACTS AND LOCATIONS:
Overall Officials: Bruce W Bode, MD, Principal Investigator — Atlanta Diabetes Associates
Locations (1):
- Atlanta Diabetes Associates, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No